CLINICAL TRIAL: NCT06220786
Title: Prospective Double Blind Controlled Trial of Low Level Laser Therapy - Cesarean Section or Vaginal Tear or Episiotomy
Brief Title: Low Level Laser Therapy for Better Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Elisabethen Krankenhaus Frankfurt GmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. Joscha Reinhard, Specialist registrar, St. Elisabethen Krankenhaus Frankfurt GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FLaser
Record Dates: First submitted 2023-12-19; First posted 2024-01-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Surgical Scar Tissue of Cesarean Section or Vaginal Tear or Episiotomy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized double blind study. Intervention 1: Low-level laser therapy ca. 72 Joules vs. Intervention 2: No Low-level laser therapy.
  Doctors & Patients do not kown which laser is the "true" laser or the "fake" laser
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding of the two laser pens is in place till all patient data has been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-level laser therapy (Active Comparator): Laser pen with low-level laser therapy.
  Interventions: Device: Low-level laser therapy
- Sham no low-level laser therapy (Sham Comparator): Identical laser pen without the low-level laser production.
  Interventions: Device: "Fake" low-level laser therapy

INTERVENTIONS:
Device: Low-level laser therapy — Low-level laser therapy ca. 72 Joules per cm2
  Arms: Low-level laser therapy
Device: "Fake" low-level laser therapy — Identical laser pen without production of low-level laser therapy
  Arms: Sham no low-level laser therapy

SUMMARY:
Prospective randomized double blind study. Intervention 1: Low-level laser therapy ca. 72 Joules vs. Intervention 2: No Low-level laser therapy.

Outcome: Pain score & would healing at discharge, 1 months & 3 months

DETAILED DESCRIPTION:
After surgical suture application of low level laser therapy of ca. 72 Joules / cm2.

Evaluation at discharge, after 1 months & 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Caesarean section or perineal tear grade 1-4 or episiotomy
* competent in German language

Exclusion Criteria:

* no caesarean section or birth without perineal tear grad 1-4 / episiotomy
* No consent given

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | Questionnaire 3 to 4 days after birth, after 1 month after birth & after 3 months after birth
  Visual analog scale (1= no pain; 10 = severe pain)

SECONDARY OUTCOMES:
subjective would healing | Questionnaire 3 to 4 days after birth, after 1 month after birth & after 3 months after birth
  Visual analog scale (1= very good healing; 10 = very bad would healing)

CONTACTS AND LOCATIONS:
Overall Officials: Joscha Reinhard, Prof. Dr., Principal Investigator — St. Elisabethenkrankenhaus Frankfurt
Locations (1):
- Prof. Dr. Joscha Reinhard, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No